CLINICAL TRIAL: NCT02801136
Title: Treatment Outcomes of Retraining and Control Therapy (ReACT) for Psychogenic Non-epileptic Seizures (PNES)
Brief Title: Treatment Outcomes of ReACT for PNES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Aaron Fobian, Principal investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F151001004
Record Dates: First submitted 2016-06-11; First posted 2016-06-15 (Estimated); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Convulsion, Non-Epileptic
MeSH Terms: conditions — Seizures | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ReACT for PNES (Experimental): ReACT consists of 8 weekly sessions of therapy focused on teaching adolescents to regain control of their body through managing thoughts and behaviors that reinforce the PNES and return to previous activities. It teaches parents how to respond to PNES in a manner that encourages the adolescents to regain control of their body. The PNES is explained as behaviors learned through classical and operant conditioning .
  Interventions: Behavioral: ReACT
- Supportive Therapy (Active Comparator): The supportive therapy treatment consists of 8 weekly sessions of therapy focused on discussing daily difficulties and/or stressors they experience and identifying stress triggers for PNES. The PNES is explained as physical manifestations of psychological stress.
  Interventions: Behavioral: Supportive Therapy
- Healthy Control (No Intervention): Healthy controls are matched to patients with PNES based on age (+ or - 1 year), gender, race and family income. They come to one laboratory visit to complete initial visit questionnaires and computer tasks.

INTERVENTIONS:
Behavioral: ReACT
  Other Names: Retraining and Control Therapy
  Arms: ReACT for PNES
Behavioral: Supportive Therapy
  Arms: Supportive Therapy

SUMMARY:
This research study is examining the effects of Retraining and Control Therapy (ReACT; an intervention focused on changing behaviors and thoughts) for psychogenic non-epileptic seizures (PNES, episodes resembling epileptic seizures but with no medical explanation). Participants engage in 8 individual therapy sessions consisting of either cognitive behavioral therapy or supportive therapy. Healthy control participants also complete pre-questionnaires and two computer tasks.

DETAILED DESCRIPTION:
Participants come to our laboratory for a total of 11 sessions. During the initial visit, participants complete several questionnaires assessing demographics, personality style, relationships with friends and family, as well as past and current PNES symptoms. They also completed two computer tasks: the magic and turbulence task and a modified Stroop task. Participants must provide EEG results indicating a diagnosis of psychogenic non-epileptic seizures.

Participants receive a PNES diary to record all episodes during the course of the study. They are randomly assigned to either receive ReACT for PNES or supportive therapy, and they return 8 times over the next 8 weeks for therapy sessions. If randomized to ReACT, participants and a family member learn how to change behaviors and thoughts to address PNES. If randomized to supportive therapy, they discuss stressors and how they relate to the PNES.

Procedures are the same for each therapy group. The first therapy session lasts approximately 90 minutes. All subsequent sessions last about one hour. After completing the 8 therapy sessions participants return one week later for a follow-up visit lasting approximately one hour. This visit consists of answering several questionnaires and an interview about current PNES symptoms. Participants return two months later for a final follow-up visit similar to the one week follow up visit. Lastly, participants and their parent are called 1 year after completing treatment and are asked to report PNES frequency over the last 30 days. They are also asked if they think ReACT was helpful, and if so, what the most helpful part of ReACT was.

Healthy controls are matched to participants with PNES based on age (+ or - 1 year), gender, race and family income. They come for 1 laboratory visit to complete the initial visit questionnaires and computer tasks.

ELIGIBILITY:
Inclusion Criteria:

* 9-18 years old.
* Diagnosis of psychogenic non-epileptic seizures by a medical doctor using video/EEG.
* Family member (parent if a minor) willing to participate and that the subject with PNES chooses.

Exclusion Criteria:

* Substance use.
* Psychosis.
* Severe intellectual disability
* Diagnosis of epilepsy is acceptable as long as patient's neurologist confirms that epileptic seizures are currently under control.

Healthy controls are matched on age (+ or - 1 year), sex, race and family income and can have no psychiatric or medical diagnosis.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 94 (Actual)
Dates: Start 2016-06; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
PNES Frequency | 14 months (4 months from baseline to 2 months after the final therapy session and then again for 30 days at the 1-year followup)
  Measured by Psychogenic Non-epileptic Seizures (PNES) diary including frequency, premonitory symptoms, description of PNES symptoms and duration. Assessed at baseline visit, 7 days after final therapy session, and 2 months after final therapy session (about 4 months total).
Stroop Task | 4 months
  Measure of cognitive inhibition and selective attention, higher scores means poorer cognitive inhibition and selective attention. Assessed at baseline visit, 7 days after final therapy session, and 2 months after final therapy session (about 4 months total).
Magic and turbulence task | 4 months
  Measure of perceived sense of control in response to tasks in which control is manipulated; Greater negative numbers indicate improved understanding of control. Assessed at baseline visit, 7 days after final therapy session, and 2 months after final therapy session (about 4 months total).

SECONDARY OUTCOMES:
Coping Skills | 4 months
  Adolescent Coping Orientation for Problem Experiences (A-Cope) will be assessed at baseline visit, 7 days after final therapy session, and 2 months after final therapy session (about 4 months total). Scores range from 54-270.
Behavior Assessment System for Children, Second Edition | 4 months
  Anxiety, Depression, Social Stress, Somatization, Relations with Parents higher scores indicate greater anxiety and depression. Scores range from 0-100. Assessed at baseline visit, 7 days after final therapy session, and 2 months after final therapy session (about 4 months total).
Pediatric Quality of Life Inventory Generic Core | 4 months
  Pediatric quality of life, greater scores indicate greater quality of life. Scores range from 0-100. Assessed at baseline visit, 7 days after final therapy session, and 2 months after final therapy session (about 4 months total).
Children's Somatic Symptoms Inventory (CSSI-24) | 4 months
  general somatic symptom complaints, higher scores indicate greater somatic complaints. Scores range from 0-140. Assessed at baseline visit, 7 days after final therapy session, and 2 months after final therapy session (about 4 months total).
Childhood Trauma Questionnaire | At baseline
  History of physical, sexual and/or emotional abuse and physical and emotional neglect, higher scores indicate greater abuse/neglect
Multidimensional Assessment of Interoceptive Awareness (MAIA) | 4 months
  Measure of components of interoceptive awareness; higher scores indicate greater presence of interoceptive awareness. Assessed at baseline visit, 7 days after final therapy session, and 2 months after final therapy session (about 4 months total).
Millon Adolescent Clinical Inventory (MACI) | At baseline
  Assesses mental health and behavior concerns in adolescents; higher scores indicate greater presence of subscale
Shipley | At baseline
  Assesses verbal IQ; higher scores indicate greater verbal IQ
Opinion of ReACT | 12 months after the final therapy session
  Parents and children are called and asked to independently report if they believed ReACT helpful and if so, what the most helpful part was.

CONTACTS AND LOCATIONS:
Locations (1):
- Sparks Center Office of Psychiatric Research, Birmingham, Alabama, United States